CLINICAL TRIAL: NCT01635322
Title: The Relationship Between Sagittal Plane Correction and Quality of Life in Adult Deformity Patients Treated With Posterior Instrumentation
Brief Title: Sagittal Plane Correction With Pass-LP Device in Adult Deformity Patients
Status: Completed | Type: Observational
Sponsor: Medicrea International (Industry)
Responsible Party: Sponsor
Other Study IDs: 0309
Record Dates: First submitted 2012-03-01; First posted 2012-07-09 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Lumbar or Thoraco-lumbar Adult Deformity
Keywords: deformity; adult; lumbar; thoraco-lumbar; Sagittal vertebral Alignement (SVA); Oswestry Disability Index (ODI)
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lumbar or thoraco-lumbar Adult Deformity: Lumbar or thoraco-lumbar Adult Deformity
  Interventions: Device: Polyaxial posterior spinal fusion system

INTERVENTIONS:
Device: Polyaxial posterior spinal fusion system — posterior correction and fusion of the thoraco-lumbar or lumbar spine
  Other Names: PASS® LP system

SUMMARY:
The purpose of this study is to evaluate the correlation between the restoration of the sagittal balance and the improvement of the Quality of Life for patients with adult scoliosis, treated with a polyaxial system (PASS® LP system) during the 2 years after a spinal fusion surgery.

ELIGIBILITY:
Inclusion criteria

* Lumbar or thoraco-lumbar Adult Deformity requiring posterior spinal instrumentation and fusion like:

  * Scoliosis
  * Kyphosis
  * Kyphoscoliosis
* Patient with a Cobb angle ≥ 30° and/or confirmed sagittal imbalance defined as sagittal vertical axis (SVA) more or equal to 5cm and/or a loss of lumbar lordosis versus the pelvic incidence
* Patient ≥ 21 years old
* Surgery that requires 4 or more levels to be operated
* Patient with complete pre-operative radiographic data: antero-posterior and lateral standing full spine x-rays (from hips to C2) and lateral bending x-rays (standing)
* Patient able to complete a self-administered questionnaire
* Patient able to sign a consent form

Exclusion criteria

* Patient operated with posterior spinal fusion without PASS LP device
* Patients who required a Vertebral Column Resection technique surgery
* Neuromuscular scoliosis or diseases and any neuro-related pathology
* Spinal cord abnormalities with any neurologic symptoms or signs
* Primary abnormalities of bones (e.g. osteogenesis imperfecta)
* Recent significant trauma
* Patient is involved in current medical litigation
* Metabolic spinal pathology
* Pathologic obesity (BMI > 40)
* Patients with infection (in particularly osteomyelitis)
* Patient < 21 years old
* Pregnancy or intended to get pregnant during the next 3 years
* Insulin-dependent diabetes
* All other contra-indications given in the PASS® LP System instructions for use
* Patient unable to sign an informed consent form
* Patient unable to complete a self-administered questionnaire

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with a lumbar or thoraco-lumbar spine deformity
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Correlation between correction of SVA and improvement ODI | preop, 3 months, 6 months, 12 months, 24 months
  The primary objective is to evaluate the correlation between:
  * the correction of the Sagittal Vertical Alignement (SVA), expressed in centimeters - SVA is the distance between C7 plumbline and the posterior of the superior endplate of S1)
  * the improvement of the Oswestry Disability Index (ODI) is the positive difference of the preoperative score and the postoperative score - expressed in % or a score (/50)

SECONDARY OUTCOMES:
Correction of the sagittal parameters | preop, 24 months
  Sagittal parameters are evaluated by:
  - Cobb angle: Thoracic kyphosis measured from T5 to T12 and between the 2 inflexion points of the curve Lumbar lordosis measured from T12 to S1 and between the 2 inflexion points of the curve
  * Pelvic Incidence (PI)
  * Pelvic Tilt (PT)
  * Sacral Slope (SS)
  * Proximal junction Cobb angle
  * T1 spinopelvic inclination (T1-SPI)
improvement of Quality of life | preop, 3 months, 6 months, 12 months, 24 months
  * The effect that the patient's pathology has on his/her daily life evaluated by the Scoliosis Research Society (SRS-22) questionnaire designed and recommended by the Scoliosis Research Society
  * Pain reduction for back and leg by the Visual Analogue Scale (VAS)
  * Patient satisfaction with the results of their operation using a simple questionnaire (Patient Satisfaction Index - PSI) which was designed and recommended by the North American Spine Society (NASS)
Complications associated with the device | preop, 3 months, 6 months, 12 months, 24 months
  Per and Post-operative device complications:
  Screw pull-out Loosening, breakage and pseudarthrosis based on x-rays analysis
Complications associated with the surgery | preop, 3 months, 6 months, 12 months, 24 months
  Peri-operative data: length of operative time, length of correction time, blood loss … Surgical complications
Coronal correction | preop, 3 months, 6 months, 12 months, 24 months
  * A pre/post-operative comparison of regular Cobb angles
  * A pre/post-operative comparison of C7 plumb line (Coronal balance)
  * A pre/post-operative comparison of Apical Vertebra Translation (AVT)
Vertebra rotation | preop, 24 months
  * A pre/post-operative comparison of Rotary Vertebra Subluxation (olisthesis)
  * A pre/post-operative comparison of Apical Vertebra Rotation (AVR) - Nash Moe
Adjacent levels degeneration | preop, 24 months
  preoperative and post-operative comparison of the disc height of the upper and lower adjacent levels
Fusion | preop, 24 months
  standing X-Rays observations (osseous formation)

CONTACTS AND LOCATIONS:
Overall Officials: Evalina BURGER, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- UC Denver, Denver, Colorado, United States
- Santy orthopedic center, Lyon, France